CLINICAL TRIAL: NCT03973528
Title: A Preliminary Evaluation of the Efficacy of Traditional Chinese Medicine in Treating Elderly Women With Infertility
Brief Title: Primary Efficacy Evaluation of Traditional Chinese Medicine in Treating Older Infertile Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201702097A3; Chang Gung MH (Other Grant/Funding Number: CMRPG3H1931)
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Infertility, Female
Keywords: anti-Mullerian hormone (AMH); Traditional Chinese Medicine(TCM); Infertility
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional Chinese medicine (Experimental): The experimental group use traditional Chinese medicine
  Interventions: Drug: traditional Chinese medicine: tonifying kidney Wan
- non- traditional Chinese medicine (No Intervention): The no intervention group no use traditional Chinese medicine.

INTERVENTIONS:
Drug: traditional Chinese medicine: tonifying kidney Wan — traditional Chinese medicine : tonifying kidney Wan
  Other Names: tonifying kidney Wan I: Zuo Gui Wan; tonifying kidney Wan II :Guilu Erxian
  Arms: traditional Chinese medicine

SUMMARY:
This study is a preliminary evaluation of the efficacy of traditional Chinese medicine in the treatment of elderly infertile women.

DETAILED DESCRIPTION:
Research design: initial acceptance of 60 people, 30 in the no intervention group and 30 in the experimental group.

The no intervention group no use Traditional Chinese medicine. The experimental group use Traditional Chinese medicine. Affect natural pregnancy and IVF success factors, the quality of ovarian function plays a very important role. Currently used to predict ovarian follicle inventory indicators, including: age, the total number of small sized ovarian follicles, the first three days of menstrual follicle-stimulating hormone, Anti-Mullerian hormone, inhibin-B.

Research Analysis Chang Gung Memorial Hospital infertility patients using traditional Chinese medicine, more than 40-year-old infertility patients, the most commonly used compound is Zuo Gui Wan. Chinese medicine believes that elderly women with infertility ovulation poor, the main pathogenesis of kidney deficiency. The proportion of domestic infertility patients has increased year by year. Traditional Chinese medicine had become popular and acceptable, but the substantial evidence and treatment consensus of infertility are scanty.

Due to the outbreak of the new crown pneumonia epidemic, which made it difficult to accept the case. Only 17 subjects in the experimental group completed the test. The average age of the subjects was 40.11 ±3.09 years old, and 9 of them were over 40 years old. The AMH before the test was all below 1.2. After three months of treatment with traditional Chinese medicine, 16 subjects had an increase in the number of small sized ovarian follicles. The average total number of small ovarian follicles before the test was 3.06±0.90, and the average increased to 4.53±1.46 after treatment. (P<0.05), which was statistically significant. Eleven subjects showed a decrease in follicle-stimulating hormone on the third day of menstruation after treatment, 9 subjects showed an increase in anti-Mullerian hormone (AMH) value after treatment, and 3 subjects had anti-Mullerian hormone (AMH) values higher than 1.2 after treatment, but they did not reach statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* A. Women aged 35-45, married, without contraception, after 12 months of normal sexual life, did not take any contraceptive measures, and did not successfully conceive women.

B. Blood tests for serum anti-Mullerian hormone ( AMH) less than 1.2, female hormones FSH, LH, E2 blood test is normal.

C. Women who are not planning for IUI or IVF in the next three months. D. Menstrual cycle rules 21-35 days. E. Willing to sign a written consent form.

Exclusion Criteria:

A. Women with contraceptive. B. Vegetarians or have been taking Traditional Chinese medicine allergies. C. The following diseases have occurred in the past six months: cancer, high blood pressure, diabetes, heart disease, stroke, myocardial infarction, hyperthyroidism or hypothyroidism, chronic hepatitis, gastric ulcer, stomach bleeding, chronic constipation or diarrhea, major trauma and surgery, severe uterine and pelvic infections.

D. Because of the need for disease, it is currently necessary to take western medicine for more than three months.

E. Women with abnormal liver function (GOT, GPT greater than 2 times the upper limit of normal).

F. Women with abnormal renal function (serum creatinine > 1.5 mg/dl). G. Poor compliance with medication. H. In the past month, take a Traditional Chinese medicine to treat infertility. I. Take DHEA for the past month.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Evaluation of Traditional Chinese medicine treatment of infertile women older than 35 years of efficacy.
Enrollment: 17 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
serum anti-Mullerian hormone (AMH) index | three months
  The efficacy of traditional Chinese medicine in the treatment of infertile women was evaluated by examining serum anti-Mullerian hormone (AMH) index
total number of small ovarian follicles by the ultrasound examination (menstrual cramps 3-5 days). | three months
  The efficacy of traditional Chinese medicine in the treatment of infertile women was evaluated by the total number of small ovarian follicles by the ultrasound examination (menstrual cramps 3-5 days).

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Tang Hsieh, MD, Study Chair — Chang Gung MH IRB
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan